CLINICAL TRIAL: NCT00537121
Title: Phase I Study of Vorinostat [Suberoylanilide Hydroxamic Acid (VORINOSTAT)] With Irinotecan, 5-Fluorouracil (5-FU) and Leucovorin (FOLFIRI) for Advanced Upper Gastrointestinal Cancers
Brief Title: Vorinostat, Irinotecan, Fluorouracil, and Leucovorin in Treating Patients With Advanced Upper Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564857; RPCI-I-78806
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer; Gastric Cancer; Liver Cancer
Keywords: recurrent gastric cancer; stage IV gastric cancer; recurrent esophageal cancer; stage IV esophageal cancer; adenocarcinoma of the esophagus; adenocarcinoma of the stomach; squamous cell carcinoma of the esophagus; adult primary hepatocellular carcinoma; stage III gastric cancer; stage III esophageal cancer; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Carcinoma, Hepatocellular | interventions — Fluorouracil; Irinotecan; Leucovorin; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
Drug: vorinostat — Taken Orally
Other: pharmacological study — Correlative Study

SUMMARY:
RATIONALE: Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as irinotecan, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat when given together with irinotecan, fluorouracil, and leucovorin in treating patients with advanced upper gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) and recommended phase II dose (RPTD) of vorinostat (SAHA) when administered continuously with standard doses of irinotecan hydrochloride, fluorouracil, and leucovorin calcium (FOLFIRI) in patients with advanced upper gastrointestinal cancer.
* Determine the MTD and RPTD of SAHA when administered intermittently with standard doses of FOLFIRI in these patients.

Secondary

* Describe the toxicity of the SAHA and FOLFIRI combination.
* Explore the effects of SAHA and FOLFIRI combination on TGF-β expression.
* Explore the alteration of survivin expression by the SAHA and FOLFIRI combination.
* Describe the effect of FOLFIRI on the pharmacokinetics of SAHA.
* Describe the effect of SAHA on the pharmacokinetics of irinotecan.
* Describe the response rate, progression-free survival, and overall survival of patients treated with this regimen.

OUTLINE: Patients receive irinotecan hydrochloride IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2 (FOLFIRI). Patients also receive oral vorinostat (SAHA) according to 1 of the following dosing regimens outlined below, depending upon time of study entry:

* Determination of maximum tolerated dose (MTD) for continuous SAHA dosing: Patients receive SAHA once daily on days 2-14 of course 1 and then on days 1-14 of all subsequent courses.
* Evaluation of SAHA pharmacokinetics at MTD for continuous dose SAHA: Patients receive SAHA on day -7 (before beginning course 1) and then once daily on days 1-14 at the MTD.
* Determination of MTD for intermittent SAHA: Patients receive SAHA once daily on days 1-7 at the MTD determined for continuous SAHA dosing. Patients receive escalating doses of SAHA until the MTD of intermittent SAHA is determined.

Treatment with FOLFIRI and vorinostat repeats every 2 weeks for 24 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo tumor tissue and blood sample collection periodically for pharmacokinetic and correlative studies. Tumor tissue samples are assessed for TGF-β expression by immunohistochemical methods and by reverse transcriptase-polymerase chain reaction for mRNA expression. Immunohistochemistry and immunoenzymatic techniques are performed to study survivin expression before beginning treatment and after completion of course 1. Pharmacokinetic studies for irinotecan, SN38, and SN38G are obtained on days 1 (before SAHA) and 15 (after SAHA). Blood is also collected for analysis of UGT1A1 polymorphism. Other patients undergo blood collection on days -7 (before FOLFIRI) and 2 (with FOLFIRI) for vorinostat Pharmacokinetic studies. Samples are analyzed by liquid chromatography-mass spectrometry.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed upper gastrointestinal tract cancer, including any of the following:

  * Esophageal cancer (adenocarcinoma or squamous cell carcinoma)
  * Gastric cancer (adenocarcinoma or squamous cell carcinoma)
  * Hepatocellular carcinoma
* Locally advanced, inoperable disease or metastatic disease
* No uncontrolled brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 (Karnofsky PS ≥ 70%)
* Life expectancy > 12 weeks
* Platelet count ≥ 100,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Leukocytes ≥ 3,000/mcL
* Total bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to understand and willing to sign a written informed consent document
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat (SAHA) or other agents used in the study
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Uncontrolled hypertension
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No coagulopathy or bleeding disorder
* No known UGT1A1 polymorphism

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy for metastatic disease
* No prior histone deacetylase inhibitors
* No concurrent prophylactic hematologic growth factors
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent valproic acid
* No other concurrent investigational therapy
* Concurrent therapeutic anticoagulation therapy is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-11; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of vorinostat (SAHA) when administered continuously and intermittently with standard doses of irinotecan hydrochloride, fluorouracil, and leucovorin calcium (FOLFIRI) | 4 weeks
Recommended phase II dose (RPTD) of SAHA when administered continuously and intermittently with standard doses of FOLFIRI | 4 weeks

SECONDARY OUTCOMES:
Toxicity of the SAHA and FOLFIRI combination | Baseline and after 2 weeks of Treatment
Effects of SAHA and FOLFIRI combination on TGF-β signaling and survivin expression | Every 6 months
Response rate | Every 6 months
Progression-free survival | Every 6 months
Overall survival | Every 3 months for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States